CLINICAL TRIAL: NCT03845296
Title: A Phase II Study of Rucaparib in Patients With Genomic LOH High and/or Deleterious BRCA1/2 Mutation Stage IV or Recurrent Non-Small Cell Lung Cancer (LUNG-MAP Sub-Study)
Brief Title: Rucaparib in Treating Patients With Genomic LOH High and/or Deleterious BRCA1/2 Mutation Stage IV or Recurrent Non-small Cell Lung Cancer (A Lung-MAP Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1900A; NCI-2018-02129 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900A (Other: SWOG); S1900A (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Deleterious BRCA1 Gene Mutation; Deleterious BRCA2 Gene Mutation; Loss of Heterozygosity; Lung Non-Small Cell Squamous Carcinoma; Recurrent Large Cell Lung Carcinoma; Recurrent Lung Adenocarcinoma; Recurrent Lung Non-Small Cell Carcinoma; Recurrent Non-Squamous Non-Small Cell Lung Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (rucaparib) (Experimental): Patients receive rucaparib PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Given PO
  Other Names: 6H-Pyrrolo(4,3,2-ef)(2)benzazepin-6-one, 8-Fluoro-1,3,4,5-tetrahydro-2-(4-((methylamino)methyl)phenyl)-; 8-Fluoro-2-(4-((methylamino)methyl)phenyl)-1,3,4,5-tetrahydro-6H-azepino(5,4,3-cd)indol-6-one

SUMMARY:
This phase II Lung-MAP trial studies how well rucaparib works in treating patients with genomic loss of heterozygosity (LOH) high and/or deleterious BRCA1/2 mutation stage IV non-small cell lung cancer or that has come back. Rucaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) (confirmed and unconfirmed, complete and partial) associated with rucaparib in patients with genomic LOH high and/or deleterious BRCA1/2 mutations within: Cohort 1: Patients with squamous cell histology or mixed histology with a squamous component; Cohort 2: Patients with non-squamous histology (adenocarcinoma, large cell, or non-small cell lung cancer [NSCLC] not otherwise specified [NOS]).

SECONDARY OBJECTIVES:

I. To evaluate investigator assessed progression-free survival (IA-PFS) and overall survival (OS) associated with rucaparib within each cohort.

II. To evaluate duration of response among responders within each cohort. III. To evaluate the frequency and severity of toxicities associated with rucaparib among all patients enrolled on the study (combining cohorts).

TRANSLATIOAL MEDICINE OBJECTIVES:

I. To evaluate the association between alterations in deoxyribonucleic acid (DNA) repair genes and response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To perform comprehensive next-generation sequencing of circulating tumor DNA (ctDNA) at baseline in all patients to assess its clinical utility in comparison to tumor tissue biomarker profiles.

III. To establish a tissue/blood repository from patients with refractory non-small cell lung cancer (NSCLC).

OUTLINE:

Patients receive rucaparib orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all SCREENING/PRE-SCREENING and SUB-STUDY REGISTRATION COMMON ELIGIBILITY CRITERIA as specified in S1400: Phase II/III Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer (Lung-Map)
* Patients must be assigned to S1900A. S1900A biomarker eligibility defined as LOH high and/or deleterious BRCA1/2 mutation is as follows using the Foundation Medicine Inc (FMI) tissue- assay:

  * LOH; alteration type: loss of heterozygosity (LOH); eligible alteration: Genomic LOH >= 21%
  * BRCA; alteration type: homologous recombination deficiency (HRD); eligible alteration: Deleterious mutations in BRCA1 or BRCA2
* Patients must not have had prior treatment with any PARP inhibitor, including rucaparib, talazoparib, veliparib, olaparib, or niraparib. For information and a list of PARP inhibitors, please consult the S1900A ? Poly Polymerase Inhibitors, Scott et al., 2015 JCO ref from the link on the S1900A protocol abstract page of the SWOG (http://swog.org) or CTSU (https://www.ctsu.org) websites.
* Patients must be able to take oral medications.
* Patients must not have a >= Grade 3 hypercholesterolaemia (defined by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) within 28 days prior to sub-study registration.
* Patients must not have EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, ROS 1 gene rearrangement, and BRAF V600E mutation unless they have progressed following all standard of care targeted therapy.
* Patients must not have documented evidence of acute hepatitis or have an active or uncontrolled infection.
* Patients with a known history of human immunodeficiency virus (HIV) seropositivity:

  * Must have undetectable viral load using standard HIV assays in clinical practice.
  * Must have CD4 count >= 400/mcL.
  * Must not require prophylaxis for any opportunistic infections (i.e., fungal, mycobacterium avium complex [mAC], or pneumocystis pneumonia [PCP] prophylaxis).
  * Must not be newly diagnosed within 12 months prior to sub-study registration.
* Patients must have progressed (in the opinion of the treating physician) following the most recent line of therapy.
* Patients must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study registration. Patients must have recovered (=< Grade 1) from any side effects of prior therapy. Patients must not have received any radiation therapy within 14 days prior to sub-study registration.
* Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
* Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to sub-study registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration. CT and MRI scans must be submitted for central review via TRIAD.
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study registration. Patient must not have leptomeningeal disease, spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to registration, AND (2) patient has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to sub-study registration.
* Patient must not have had a major surgery within 14 days prior to sub-study registration. Patient must have fully recovered from the effects of prior surgery in the opinion of the treating investigator.
* Absolute neutrophil count (ANC) >= 1,500/mcl (obtained within 28 days prior to sub-study registration)
* Platelet count >= 100,000 mcl (obtained within 28 days prior to sub-study registration)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to sub-study registration)
* Serum bilirubin =< Institutional Upper Limit of Normal (IULN). For patients with liver metastases, bilirubin must be =< 5 x IULN (within 28 days prior to sub-study registration)
* Either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN (if both ALT and AST are done, both must be < 2 IULN). For patients with liver metastases, either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN) (within 28 days prior to sub-study registration)
* Patients must have a serum creatinine =< the IULN OR calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to sub-study registration.
* Patients must have Zubrod performance status 0-1 documented within 28 days prior to sub-study registration.
* Patients must not have any Grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia.
* Pre-study history and physical exam must be obtained within 28 days prior to sub-study registration.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.
* Patients must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method during the study and 6 months after study completion. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures during the study and 6 months after study completion
* Patients must agree to have blood specimens submitted for circulating tumor DNA (ctDNA).
* Patients must also be offered participation in banking and in the correlative studies for collection and future use of specimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Riess, Principal Investigator — SWOG Cancer Research Network
Locations (950):
- United States (950):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Hematology Oncology Consultants Limited-Darien, Darien, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Loyola Center for Cancer Care and Research, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Saint Claire Regional Medical Center, Morehead, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - University of Rochester, Rochester, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Rex Hematology Oncology Associates-Cary, Cary, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Hematology Oncology Associates-Garner, Garner, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Saint Clair Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 64 participants were initially enrolled. Three participants were ineligible, one was not analyzable and one withdrew consent prior to starting the study drug. In all, 59 participants were eligible and included in the analysis: 25 in the squamous cohort and 34 in the non-squamous cohort.
Groups:
- Cohort 1: Squamous: Participants with squamous cell lung cancer
- Cohort 2: Non-Squamous: Participants with non-squamous cell lung cancer (adenocarcinoma, large cell, NSCLC NOS, mixed histology with any non-squamous component)
Period: Overall Study
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous
Started | 25 | 34
Completed | 0 | 0
Not Completed | 25 | 34
Not completed — On Treatment | 2 | 1
Not completed — Adverse Event | 4 | 11
Not completed — Refusal unrelated to adverse event | 0 | 1
Not completed — Progression/relapse | 14 | 18
Not completed — Death | 4 | 0
Not completed — Other - not protocol specified | 1 | 3

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous | Total
Number analyzed (Participants) | 25 | 34 | 59
Age, Continuous [Median (Full Range); unit: years] | 63.9 [48.1 to 83.6] | 69.1 [54.0 to 82.3] | 65.7 [48.1 to 83.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 33 | 58
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 23 | 30 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Prior Lines of Treatment for Stage IV Disease [Count of Participants; unit: Participants]
  0 | 1 | 0 | 1
  1 | 9 | 16 | 25
  2 or more | 15 | 18 | 33
Performance Status [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status Scale:
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 4 | 11 | 15
    1 | 21 | 23 | 44
Weight Loss in the Past 6 Months [Count of Participants; unit: Participants]
  < 5% | 16 | 24 | 40
  5 - < 10% | 5 | 6 | 11
  10 - < 20% | 3 | 3 | 6
  >= 20% | 0 | 1 | 1
  Unknown | 1 | 0 | 1
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 10 | 10 | 20
  Former Smoker | 15 | 20 | 35
  Never Smoker | 0 | 4 | 4
Study Biomarker Status [Count of Participants; unit: Participants]
  LOH Only | 16 | 20 | 36
  LOH and BRCA1 | 1 | 3 | 4
  LOH and BRCA2 | 3 | 1 | 4
  BRCA1 Only | 0 | 4 | 4
  BRCA2 Only | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Percentage of participants with a complete or partial, confirmed or unconfirmed response.
  Complete Response (CR): Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  Partial Response (PR): Applies only to participants with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous
Number analyzed (Participants) | 25 | 34
Percentage of participants | 8 [0 to 19] | 12 [1 to 23]

2. Secondary Outcome: Investigator-Assessed Progression-Free Survival (IA-PFS)
Description: Time from date of registration to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan (as defined by the disease assessment schedule) is used as the date of progression.
  Progression: One or more of: 20% increase in sum of diameters of target lesions over smallest sum observed and absolute increase of at least 0.5cm; Unequivocal progression of non-measurable disease in opinion of the treating physician; Appearance of any new lesion/site; Death due to disease w/o prior progression or symptomatic deterioration Symptomatic deterioration: Global deterioration of health status requiring treatment discontinuation w/o objective evidence of progression
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous
Number analyzed (Participants) | 25 | 34
months | 2.9 [1.6 to 6.2] | 3.5 [1.6 to 4.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Time from date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous
Number analyzed (Participants) | 25 | 34
months | 8.2 [4.4 to 15.3] | 7.8 [5.0 to 11.4]

4. Secondary Outcome: Duration of Response (DoR)
Description: Time from date of first documentation of response (complete or partial) to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause among participants who achieve a response. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan will be used as the date of progression.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants who had a response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Squamous | Cohort 2: Non-Squamous
Number analyzed (Participants) | 2 | 4
months | NA [NA to NA] — Median not reached | 14.9 [9.9 to NA] — Insufficient follow-up data

5. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 5.0 was used for routine toxicity reporting and serious adverse events (SAEs).
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Eligible participants who received at least one dose of protocol treatment
Measure: Number; unit: Participants
Groups:
- Rucaparib: Participants receive rucaparib PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Rucaparib
Number analyzed (Participants) | 59
Participants
  Alanine aminotransferase increased | 2
  Alkaline phosphatase increased | 1
  Anemia | 13
  Aspartate aminotransferase increased | 1
  Blood bilirubin increased | 1
  Chronic kidney disease | 1
  Confusion | 1
  Dyspnea | 2
  Fatigue | 5
  Generalized muscle weakness | 2
  Hypertension | 1
  Hypokalemia | 2
  Lymphocyte count decreased | 5
  Nausea | 1
  Neutrophil count decreased | 2
  Personality change | 1
  Platelet count decreased | 3
  Rash maculo-papular | 1
  Vomiting | 1
  White blood cell decreased | 3

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 3 years post registration
Description: CTCAE Version 5.0 was used for routine toxicity reporting and Serious Adverse Event (SAE) reporting. 59 participants were assessed for adverse events: 25 in the squamous cohort and 34 in the non-squamous cohort.
Arm/Group | Rucaparib
All-Cause Mortality (participants affected / at risk) | 50/59
Serious Adverse Events (participants affected / at risk) | 32/59
Other Adverse Events (participants affected / at risk) | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib (N=59)
Anemia (Blood and lymphatic system disorders) | 11
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Small intestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Disease progression (General disorders) | 4
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib (N=59)
Anemia (Blood and lymphatic system disorders) | 39
Sinus tachycardia (Cardiac disorders) | 3
Blurred vision (Eye disorders) | 5
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 14
Chills (General disorders) | 4
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 36
Fever (General disorders) | 4
Pain (General disorders) | 5
Lung infection (Infections and infestations) | 6
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 21
Alkaline phosphatase increased (Investigations) | 20
Aspartate aminotransferase increased (Investigations) | 24
Blood bilirubin increased (Investigations) | 10
Blood lactate dehydrogenase increased (Investigations) | 4
Cholesterol high (Investigations) | 15
Creatinine increased (Investigations) | 20
Investigations-Other (Investigations) | 5
Lymphocyte count decreased (Investigations) | 22
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 22
Weight loss (Investigations) | 13
White blood cell decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 22
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 16
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hot flashes (Vascular disorders) | 3
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 7
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT03845296/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT03845296/ICF_001.pdf